CLINICAL TRIAL: NCT01098032
Title: Renal Insufficiency Following Contrast Media Administration Trial II (Remedial II): The RenalGuard System in High-Risk Patients for Contrast-Induced Acute Kidney Injury
Brief Title: RenalGuard System and Contrast Media
Acronym: REMEDIALII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Carlo Briguori, MD, PhD, Clinica Mediterranea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCTCM01
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease
Keywords: Contrast media; Kidney; Complication
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic alone therapy group (Active Comparator): Systemic alone therapy group will be treated by intravenous sodium bicarbonate plus NAC administration. Patients allocated to the Systemic alone therapy group will receive 154 mEq/l of sodium bicarbonate in dextrose and H2O, according to the protocol reported by Merten et al. (9) The initial i.v. bolus was 3 ml/kg per hour for 1 hour immediately before contrast injection. Following this, patients will receive the same fluid at a rate of 1 ml/kg per hour during contrast exposure and for 6 hours after the procedure. All patients will receive NAC (Fluimucil, Zambon Group SpA, Milan, Italy) orally at a dose of 1200 mg twice daily on the day before and on the day of administration of the contrast agent (total of 2 days. Additional NAC dose (1.2 g) will be administered i.v. during the procedure.
  Interventions: Drug: Systemic alone therapy
- RenalGuard System group (Experimental): Prophylactic controlled hydration with saline (0.9%) plus N-acetylcystein (NAC; 6 g in total). In the RenalGuard group, an initial bolus (priming) of 250 ml will be administered. In case of left ventricular dysfunction (ejection fraction ≤30%) and/or unstable hemodynamic conditions the bolus will be reduced to 150 ml. Following the initial bolus, furosemide (0.25 mg/kg) will be administered in order to achieve the optimal urine flow (≥300 ml/h). The hydration will be continued throughout the duration of the procedure and will last 4 hours following the procedure. Additional doses of furosemide are allowed in case of decrease of urine flow <300 ml/h.
  Interventions: Device: RenalGuard system

INTERVENTIONS:
Device: RenalGuard system — The RenalGuard™ System (PLC Medical Systems, Inc.) is a real-time measurement and real time matched fluid replacement device designed to accommodate the RenalGuard Therapy. The RenalGuard Therapy is based on the concept demonstrated by clinical data that high urine output is beneficial to patients with impaired baseline renal function who receive intravascular iodinated contrast medio (CM). The RenalGuard System seems to be ideal for the prevention of CI-AKI, by allowing an optimal urine flow rate >300 ml/h. It is known that excessive diuresis can cause dehydration which increases the risk to the kidneys from CM. The RenalGuard System should allow the patient to achieve high urine output safely by maintaining the intravascular blood volume and avoiding the risk of over-or-under-hydration.
  Arms: RenalGuard System group
Drug: Systemic alone therapy — Patients allocated to the Systemic alone therapy group will receive 154 mEq/l of sodium bicarbonate in dextrose and H2O, according to the protocol reported by Merten et al. The initial intravenous bolus was 3 ml/kg per hour for 1 hour immediately before contrast injection. Following this, patients will receive the same fluid at a rate of 1 ml/kg per hour during contrast exposure and for 6 hours after the procedure. All patients will receive NAC (Fluimucil, Zambon Group SpA, Milan, Italy) orally at a dose of 1200 mg twice daily on the day before and on the day of administration of the contrast agent (total of 2 days)
  Other Names: Sodium Bicarbonate and N-acetylcysteine
  Arms: Systemic alone therapy group

SUMMARY:
The purpose of the present study is to assess the role of the RenalGuard System as compared to the optimal strategy (sodium bicarbonate infusion plus N-acetylcysteine (NAC)) in high and very-high risk patients to prevent contrast-induced acute kidney injury contrast induced acute kidney injury (CI-AKI).

Consecutive patients with chronic kidney disease, referred to our institutions for coronary and/or peripheral procedures, will be randomly assigned to 1) prophylactic administration of sodium bicarbonate plus NAC (Systemic alone therapy group; n > 133) and 2) RenalGuard System treatment (RenalGuard group; n > 133). All enrolled patients must have an estimated glomerular filtration rate <30 ml/min/1.73 m2 and/or a contrast nephropathy risk score ≥11). In all cases iodixanol (an iso-osmolar, non ionic contrast agent) will be administered. The primary end point is an increase of >=0.3 mg/dL in the creatinine concentration 48 hours after the procedure.

This study will give important answers on how to prevent CI-AKI in high and very-high risk patients undergoing contrast media exposure.

DETAILED DESCRIPTION:
The strategy of volume supplementation by sodium bicarbonate plus N-acetylcysteine (NAC) seems to be the optimal pharmacological approach in preventing contrast induced acute kidney injury (CI-AKI) in patients at medium-to-high risk. Whether this prophylactic strategy is effective in high and very-high risk patients is unknown. In this subset of patients the potential protective effects and therapeutic advantage of a local delivery of protective compounds should be investigated. The RenalGuard™ System (PLC Medical Systes, Inc.) is a real-time measurement and real time matched fluid replacement device designed to accommodate the RenalGuard Therapy. The RenalGuard Therapy is based on the theory that creating and maintaining a high urine output is beneficial to patients undergoing imaging procedures where contrast agents are used. This should allow the body to rapidly eliminate contrast, reducing its toxic effects. The RenalGuard System seems to be ideal for the prevention of CI-AKI, by allowing an optimal urine flow rate >150 ml/h (ideally >300 ml/h). Preliminary data suggests that the RenalGuard System, by increasing the urine flow rate ≥ 300 ml/h, allows a quick renal first-pass elimination and therefore reduces the risk for contrast nephropathy. The potential benefits of RenalGuard Therapy are intended to reduce the incidence of CI-AKI via a combination of known physiological effects of high urine output including: a) lower concentration of contrast in the kidneys, b) more rapid transit of contrast through the kidneys, c) less overall exposure to toxic contrast, d) potential reduction of oxygen consumption in the medulla of the kidneys. No randomized study has been performed to assess the role of the RenalGuard System as compared to the optimal strategy (sodium bicarbonate infusion plus NAC) in high and very-high risk patients to prevent CI-AKI.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Chronic kidney disease (estimated glomerular filtration rate <=30 ml/min/1.72 m2) and/or
3. Risk score for contrast nephropathy ≥11 (according to the Mehran score; J Am Coll Cardiol 2004; 44: 1393-1399)

Exclusion Criteria:

1. Pregnancy
2. Heart failure (NYHA functional class III-IV)
3. Acute pulmonary edema
4. Acute myocardial infarction
5. Recent (<=2 days) contrast media exposure
6. Patients enrolled in concomitant studies
7. Administration of theophylline, dopamine, mannitol and fenoldopam.
8. End-stage CKD (patients on chronic dialysis)
9. Systemic hypotension (systolic blood pressure < 100 mg/dl).
10. Multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Briguori, MD, PhD, Principal Investigator — Clinica Mediterranea, Naples,. ITALY
Locations (4):
- Italy (4):
  - Unversity of Ferrara, Department of Cardiology, Ferrara
  - IRCCS Multimedica, Milan
  - Unversity School of Medicine of Modena, Deparment of Cardiology, Modena
  - Clinica Mediterranea, Naples

REFERENCES:
- [Background] Tepel M, Aspelin P, Lameire N. Contrast-induced nephropathy: a clinical and evidence-based approach. Circulation. 2006 Apr 11;113(14):1799-806. doi: 10.1161/CIRCULATIONAHA.105.595090. No abstract available. PMID 16606801
- [Background] Gruberg L, Mehran R, Dangas G, Mintz GS, Waksman R, Kent KM, Pichard AD, Satler LF, Wu H, Leon MB. Acute renal failure requiring dialysis after percutaneous coronary interventions. Catheter Cardiovasc Interv. 2001 Apr;52(4):409-16. doi: 10.1002/ccd.1093. PMID 11285590
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Solomon R, Deray G; Consensus Panel for CIN. How to prevent contrast-induced nephropathy and manage risk patients: practical recommendations. Kidney Int Suppl. 2006 Apr;(100):S51-3. doi: 10.1038/sj.ki.5000375. No abstract available. PMID 16612402
- [Background] Persson PB, Hansell P, Liss P. Pathophysiology of contrast medium-induced nephropathy. Kidney Int. 2005 Jul;68(1):14-22. doi: 10.1111/j.1523-1755.2005.00377.x. PMID 15954892
- [Background] Tepel M, van der Giet M, Schwarzfeld C, Laufer U, Liermann D, Zidek W. Prevention of radiographic-contrast-agent-induced reductions in renal function by acetylcysteine. N Engl J Med. 2000 Jul 20;343(3):180-4. doi: 10.1056/NEJM200007203430304. PMID 10900277
- [Background] DiMari J, Megyesi J, Udvarhelyi N, Price P, Davis R, Safirstein R. N-acetyl cysteine ameliorates ischemic renal failure. Am J Physiol. 1997 Mar;272(3 Pt 2):F292-8. doi: 10.1152/ajprenal.1997.272.3.F292. PMID 9087670
- [Background] Tariq M, Morais C, Sobki S, Al Sulaiman M, Al Khader A. N-acetylcysteine attenuates cyclosporin-induced nephrotoxicity in rats. Nephrol Dial Transplant. 1999 Apr;14(4):923-9. doi: 10.1093/ndt/14.4.923. PMID 10328471
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Spargias K, Alexopoulos E, Kyrzopoulos S, Iokovis P, Greenwood DC, Manginas A, Voudris V, Pavlides G, Buller CE, Kremastinos D, Cokkinos DV. Ascorbic acid prevents contrast-mediated nephropathy in patients with renal dysfunction undergoing coronary angiography or intervention. Circulation. 2004 Nov 2;110(18):2837-42. doi: 10.1161/01.CIR.0000146396.19081.73. Epub 2004 Oct 18. PMID 15492300
- [Background] Briguori C, Airoldi F, D'Andrea D, Bonizzoni E, Morici N, Focaccio A, Michev I, Montorfano M, Carlino M, Cosgrave J, Ricciardelli B, Colombo A. Renal Insufficiency Following Contrast Media Administration Trial (REMEDIAL): a randomized comparison of 3 preventive strategies. Circulation. 2007 Mar 13;115(10):1211-7. doi: 10.1161/CIRCULATIONAHA.106.687152. Epub 2007 Feb 19. PMID 17309916
- [Background] Stone GW, McCullough PA, Tumlin JA, Lepor NE, Madyoon H, Murray P, Wang A, Chu AA, Schaer GL, Stevens M, Wilensky RL, O'Neill WW; CONTRAST Investigators. Fenoldopam mesylate for the prevention of contrast-induced nephropathy: a randomized controlled trial. JAMA. 2003 Nov 5;290(17):2284-91. doi: 10.1001/jama.290.17.2284. PMID 14600187
- [Background] McCullough PA. Contrast-induced acute kidney injury. J Am Coll Cardiol. 2008 Apr 15;51(15):1419-28. doi: 10.1016/j.jacc.2007.12.035. PMID 18402894
- [Background] Romano G, Briguori C, Quintavalle C, Zanca C, Rivera NV, Colombo A, Condorelli G. Contrast agents and renal cell apoptosis. Eur Heart J. 2008 Oct;29(20):2569-76. doi: 10.1093/eurheartj/ehn197. Epub 2008 May 8. PMID 18468994
- [Background] Stevens MA, McCullough PA, Tobin KJ, Speck JP, Westveer DC, Guido-Allen DA, Timmis GC, O'Neill WW. A prospective randomized trial of prevention measures in patients at high risk for contrast nephropathy: results of the P.R.I.N.C.E. Study. Prevention of Radiocontrast Induced Nephropathy Clinical Evaluation. J Am Coll Cardiol. 1999 Feb;33(2):403-11. doi: 10.1016/s0735-1097(98)00574-9. PMID 9973020
- [Background] Solomon R, Werner C, Mann D, D'Elia J, Silva P. Effects of saline, mannitol, and furosemide on acute decreases in renal function induced by radiocontrast agents. N Engl J Med. 1994 Nov 24;331(21):1416-20. doi: 10.1056/NEJM199411243312104. PMID 7969280
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Briguori C, Colombo A, Violante A, Balestrieri P, Manganelli F, Paolo Elia P, Golia B, Lepore S, Riviezzo G, Scarpato P, Focaccio A, Librera M, Bonizzoni E, Ricciardelli B. Standard vs double dose of N-acetylcysteine to prevent contrast agent associated nephrotoxicity. Eur Heart J. 2004 Feb;25(3):206-11. doi: 10.1016/j.ehj.2003.11.016. PMID 14972420
- [Derived] Quintavalle C, Anselmi CV, De Micco F, Roscigno G, Visconti G, Golia B, Focaccio A, Ricciardelli B, Perna E, Papa L, Donnarumma E, Condorelli G, Briguori C. Neutrophil Gelatinase-Associated Lipocalin and Contrast-Induced Acute Kidney Injury. Circ Cardiovasc Interv. 2015 Sep;8(9):e002673. doi: 10.1161/CIRCINTERVENTIONS.115.002673. PMID 26333343
- [Derived] Briguori C, Visconti G, Focaccio A, Airoldi F, Valgimigli M, Sangiorgi GM, Golia B, Ricciardelli B, Condorelli G; REMEDIAL II Investigators. Renal Insufficiency After Contrast Media Administration Trial II (REMEDIAL II): RenalGuard System in high-risk patients for contrast-induced acute kidney injury. Circulation. 2011 Sep 13;124(11):1260-9. doi: 10.1161/CIRCULATIONAHA.111.030759. Epub 2011 Aug 15. PMID 21844075
- [Derived] Briguori C, Visconti G, Ricciardelli B, Condorelli G; REMEDIAL II Investigators. Renal insufficiency following contrast media administration trial II (REMEDIAL II): RenalGuard system in high-risk patients for contrast-induced acute kidney injury: rationale and design. EuroIntervention. 2011 Apr;6(9):1117-22, 7. doi: 10.4244/EIJV6I9A194. PMID 21518686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with CKD scheduled for coronary and/or peripheral angiography/angioplasty from January 2009 to December 2011 were screened for inclusion/exclusion criteria. The trial was conducted in across 4 interventional cardiology centers in Italy, according to the principles of the Declaration of Helsinki and Good Clinical Practice
Pre-assignment Details: Two enrolled patients did not finally undergo the scheduled treatment due to the occurrence fever or gastrointestinal bleeding
Groups:
- Systemic Alone Therapy Group: Systemic alone therapy grou will be treated by intravenous sodium bicarbonate plus NAC administration. Patients allocated to the Systemic alone therapy group will receive 154 mEq/l of sodium bicarbonate in dextrose and H2O, according to the protocol reported by Merten et al. (9) The initial intravenous bolus was 3 ml/kg per hour for 1 hour immediately before contrast injection. Following this, patients will receive the same fluid at a rate of 1 ml/kg per hour during contrast exposure and for 6 hours after the procedure. All patients will receive NAC (Fluimucil, Zambon Group SpA, Milan, Italy) orally at a dose of 1200 mg twice daily on the day before and on the day of administration of the contrast agent (total of 2 days. Additional NAC dose (1.2 g) will be administered i.v. during the procedure.
Period: Overall Study
Arm/Group | Systemic Alone Therapy Group | RenalGuard System Group
Started | 147 (1 patient di not receive the treatment. Therefore this patient was excluded from the analysis.) | 147 (1 patient di not receive the treatment. Therefore this patient was excluded from the analysis.)
Completed | 146 | 146
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systemic Alone Therapy Group | RenalGuard System Group | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 14 | 33
  >=65 years | 128 | 133 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (9) | 76 (8) | 75 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 57 | 100
  Male | 104 | 90 | 194
Region of Enrollment [Number; unit: participants]
  Italy | 147 | 147 | 294

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Contrast-induced Acute Kidney Injury
Description: The primary outcome measure will be the rate of development of CI-AKI in the 2 study arms (number of participants). CI-AKI is defined as an increase in the serum creatinine concentration >=0.3 mg/dL from the baseline value at 48 hours after administration of the contrast media or the need for dialysis.
Time Frame: at 48 hours following contrast exposure
Population: all consecutive patients with chronic kidney disease scheduled for coronary and/or peripheral angiography and/or angioplasty with an estimated glomerular filtration rate (eGFR) ≤30 ml/min/1.73 m2 and/or a risk score ≥11 were considered eligible for the study
Measure: Number; unit: participants
Arm/Group | Systemic Alone Therapy Group | RenalGuard System Group
Number analyzed (Participants) | 147 | 147
participants | 146 | 146

2. Secondary Outcome: Rate of Kidney Injury and Major Adverse Events
Description: an increase in the serum creatinine concentration >=0.25% and >=0.5 mg/dl at 48 hours after contrast exposure
Time Frame: 7 days
Reporting Status: Not Posted

3. Secondary Outcome: Changes in the Serum Cystatin C Concentration at 24 and 48 Hours After Contrast Exposure
Description: Cystatin C is an alternative biomarker of kidney damage. Cystatin C seems to be superior to serum creatinine an identifying kidney function and damage.
Time Frame: 7 days
Reporting Status: Not Posted

4. Secondary Outcome: Changes in the Urine and Serum NGAL Concentration After Contrast Exposure
Description: NGAL is a new biomarker which seems to be very promising in detecting kidney injury. prelimiary data suggest that urine and serum NGAL increase very early (within few horurs) after the occurrence og acute kidney damage. Therefore, NGAL may be a real marker of acute kidney injury.
Time Frame: 7 days
Reporting Status: Not Posted

5. Secondary Outcome: the Rate of Acute Renal Failure Requiring Dialysis
Description: occurrence of renal failure requiring dialysis represents the haard endpoint of the study. Actually this represents the worst clinical consequence of CI-AKI.
Time Frame: 1 month
Reporting Status: Not Posted

6. Secondary Outcome: The Rate of In-hospital Major Adverse Events (i.e. Acute Myocardial Infarction, c) Renal Failure Requiring Dialysis, and d) Acute Pulmonary Edema)
Description: Assessment of the rate of in-hospital major adverse events (i.e. acute myocardial infarction, c) renal failure requiring dialysis, and d) acute pulmonary edema) will give important informantion on the clinical relevance of prophylactic strategies in preventing CI-AKI
Time Frame: 1 month
Reporting Status: Not Posted

7. Secondary Outcome: The Cost-effectiveness Ratio.
Description: Assessement of the cost-effectiveness ratio is important when testing a new strategy of both therapy and prophylaxis. The Renalguard system is more expensive than the conventional hydration regimen. The cost of RenalGuard system is approximately 800 $. This cost will be justified only if the system is more effective in preventing CI-AKI and improving the clinical outcome, expecially reducing the lenght of ospedalization and the rate of dialysis.
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- RenalGuard System Group: Prophylactic controlled hydration with saline (0.9%) plus N-acetylcystein (NAC; 6 g in total). In the RenalGuard group, an initial bolus (priming) of 250 ml will be administered. In case of left ventricular dysfunction (ejection fraction ≤30%) and/or unstable hemodynamic conditions the bolus will be reduced to 150 ml. Following the initial bolus, furosemide (0.25 mg/kg) will be administered in order to achieve the optimal urine flow (≥300 ml/h). The hydration will be continued throughout the duration of the procedure and will last 4 hours following the procedure.
- Systemic Alone Therapy Group: Systemic alone therapy group was treated by intravenous sodium bicarbonate plus NAC administration.
Arm/Group | RenalGuard System Group | Systemic Alone Therapy Group
Serious Adverse Events (participants affected / at risk) | 10/146 | 14/146
Other Adverse Events (participants affected / at risk) | 10/146 | 3/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RenalGuard System Group (N=146) | Systemic Alone Therapy Group (N=146)
Death (General disorders) | 6 (6) | 6 (6)
Dialysis (Renal and urinary disorders) | 1 (1) | 7 (7)
Acute pulmonary edema (Cardiac disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RenalGuard System Group (N=146) | Systemic Alone Therapy Group (N=146)
Micturation (Renal and urinary disorders) | 4 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes